CLINICAL TRIAL: NCT00005486
Title: Lymphangioleiomyomatosis (LAM) Registry
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5002; U01HL058440 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-12

CONDITIONS: Lung Diseases; Lymphangiomyomatosis
MeSH Terms: conditions — Lung Diseases; Lymphangioleiomyomatosis

SUMMARY:
To establish a registry of individuals with LAM by forming a consortium of six clinical centers and referring physicians who treat LAM patients.

DETAILED DESCRIPTION:
BACKGROUND:

LAM is a rare multi-system disease that can affect the lungs of young women, is of uncertain cause, is usually progressive, and can cause debilitating lung disease which may be corrected with lung transplantation. Several hundred women with the disease have been identified, largely through a LAM Foundation in Cincinnati, Ohio.

DESIGN NARRATIVE:

The Data and Coordinating Center is located at the Cleveland Clinic Foundation. The registry has six major clinical centers: Cleveland Clinic Foundation, Mayo Clinic-Rochester, National Heart, Lung, and Blood Institute, National Jewish Medical and Research Center, New England Medical Center, and Stanford University Medical Center. Data and lung tissue collected by the registry will be used to characterize the clinical features and natural history of the disease and to determine the efficacy of lung transplantation in this disorder. Eligible patients are to be seen yearly for up to 4 years at the Clinical Centers or, in some cases, by individual referring physicians. Tissue collected by the LAM Registry will be stored at a central NHLBI repository. Outcome events include measures of pulmonary function (eg, spirometry and, when available, lung volumes and diffusing capacity), arterial blood gases or oximetry, walking and resting oxygen titration, cardiopulmonary stress testing, cause-specific mortality, functional status, and clinical events associated with lung transplantation.

The Office of Research on Women's Health provided funding in FY 1997 in the amount of $100,000.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-07; Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Beck — The Cleveland Clinic

REFERENCES:
- [Background] Sullivan EJ, Stoller JK. The registry for individuals with lymphangioleiomyomatosis. In J. Moss, editor. LAM and Other Diseases Characterized by Smooth Muscle Proliferation. Marcel Dekker, New York, NY, pp 99-110, 1998.
- [Background] Sullivan EJ, Beck GJ, Peavy HH, Fanburg BL. Lymphangioleiomyomatosis Registry. Chest. 1999 Jan;115(1):301. doi: 10.1378/chest.115.1.301. No abstract available. PMID 9925106
- [Background] Sullivan EJ. Lymphangioleiomyomatosis: a review. Chest. 1998 Dec;114(6):1689-703. doi: 10.1378/chest.114.6.1689. No abstract available. PMID 9872207
- [Background] Ryu JH, Moss J, Beck GJ, Lee JC, Brown KK, Chapman JT, Finlay GA, Olson EJ, Ruoss SJ, Maurer JR, Raffin TA, Peavy HH, McCarthy K, Taveira-Dasilva A, McCormack FX, Avila NA, Decastro RM, Jacobs SS, Stylianou M, Fanburg BL; NHLBI LAM Registry Group. The NHLBI lymphangioleiomyomatosis registry: characteristics of 230 patients at enrollment. Am J Respir Crit Care Med. 2006 Jan 1;173(1):105-11. doi: 10.1164/rccm.200409-1298OC. Epub 2005 Oct 6. PMID 16210669